CLINICAL TRIAL: NCT07055724
Title: Exploratory Clinical Study of Fully Human BCMA Chimeric Antigen Receptor Autologous T-cell Injection (Equecabtagene Autoleucel, Eque-cel) for the Treatment of Newly Diagnosed Mayo Stage IIIb AL Amyloidosis Patients
Brief Title: Study of Eque-cel CAR-T Therapy in Newly Diagnosed Severe AL Amyloidosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Nanjing IASO Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT103ACI003
Record Dates: First submitted 2025-06-26; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: AL Amyloidosis
Keywords: Eque-cel; CAR-T; Mayo Stage IIIb
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eque-cel Arm (Experimental): Eque-cel : a dose of 1.0 x 10^6 CAR-T cells/kg
  Interventions: Biological: Eque-cel CAR-T Therapy

INTERVENTIONS:
Biological: Eque-cel CAR-T Therapy — Participants in this arm receive a single infusion of Eque-cel at a dose of 1.0 x 10^6 CAR-T cells/kg following lymphodepletion preconditioning with fludarabine and cyclophosphamide. Eque-cel is a fully human BCMA-targeted CAR-T cell therapy designed to recognize and eliminate BCMA-expressing cells.

SUMMARY:
The goal of this clinical trial is to learn if Equecabtagene Autoleucel(Eque-cel), a Chimeric Antigen Receptor T-cell (CAR-T) therapy, works to treat severe Light Chain (AL) Amyloidosis in newly diagnosed adults with Mayo Stage IIIb. It will also learn about the safety and effects of Eque-cel. The main questions it aims to answer are:

Does Eque-cel lead to hematologic remission (achieving a very good partial response or better) in AL amyloidosis? How safe is Eque-cel for these patients, and what side effects might occur?

Participants will:

Undergo blood cell collection to create personalized Eque-cel therapy. Receive pre-treatment to prepare their body for the therapy (lymphodepletion). Receive a single infusion of Eque-cel. Be monitored closely for 24 weeks after infusion, followed by long-term checkups for up to 15 years.

DETAILED DESCRIPTION:
This exploratory clinical trial investigates the efficacy and safety of Eque-cel , a fully human B-cell Maturation Antigen (BCMA)-targeted CAR-T cell therapy, in treating newly diagnosed Mayo Stage IIIb AL amyloidosis, a rare and severe systemic disorder characterized by abnormal plasma cell proliferation and amyloid fibril deposition leading to organ dysfunction. Current treatments, such as high-dose chemotherapy with stem cell transplantation or daratumumab-based regimens, fail to meet the urgent needs of Stage IIIb patients due to severe cardiac involvement, poor tolerability, and lack of approved standard therapies, necessitating rapid, low-cardiotoxicity interventions. Eque-cel, approved for relapsed/refractory multiple myeloma in China, has shown promise in prior studies with high hematologic response rates and rapid action, offering a potential solution for this high-risk population.

This study is an interventional clinical trial focused on treating newly diagnosed Mayo Stage IIIb AL Amyloidosis patients. It is a Phase II exploratory study aimed at initially validating the efficacy and safety of Eque-cel. The study employs a single-arm, open-label design, with all participants receiving Eque-cel CAR-T cell therapy (at a dose of 1.0×10⁶ CAR-T cells/kg), without randomization or blinding, to directly assess treatment outcomes. The trial is conducted at a single center (Zhongshan Hospital, Fudan University) and plans to enroll up to 17 participants. The process includes peripheral blood mononuclear cell (PBMC) collection, optional bridging therapy, lymphodepletion preconditioning, and cell infusion, followed by a 24-week primary follow-up period and long-term monitoring for up to 15 years. The study aims to complete patient enrollment within 2 years. The primary endpoint is to evaluate the hematologic response rate post-treatment, while secondary endpoints include safety and survival-related metrics. Through innovative CAR-T therapy, this study seeks to address unmet clinical needs and provide new treatment hope for this high-risk population.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged ≥18 years, regardless of gender.
2. Performance status: Eastern Cooperative Oncology Group (ECOG) performance status score ≤2.
3. Clinically diagnosed with newly diagnosed AL (light chain) amyloidosis, classified as Mayo Stage IIIb per the revised 2004 Mayo Clinic staging system at screening, with serum N-terminal pro-brain natriuretic peptide (NT-proBNP) >8500 ng/L and serum cardiac troponin T (cTnT) >0.035 μg/L or cardiac troponin I (cTnI) >0.01 g/L.
4. Presence of measurable hematologic disease at screening, defined as at least one of the following:

   1. Difference in free light chains (dFLC) >4 mg/dL, or
   2. Involved free light chain (iFLC) >4 mg/dL with abnormal kappa/lambda (κ/λ) ratio, or
   3. Serum protein electrophoresis (SPEP) M protein >0.5 g/dL.
5. Histopathological diagnosis of amyloidosis based on polarized light microscopy of Congo red-stained tissue specimens showing green birefringence, with confirmation of AL-derived amyloid deposits by at least one of the following methods:

   1. Immunohistochemistry/immunofluorescence,
   2. Mass spectrometry,
   3. Electron microscopy for characteristic appearance/immunoelectron microscopy.
6. Presence of clonal plasma cells in bone marrow, detectable by light microscopy or flow cytometry.
7. Presence of M protein in blood or urine, with exclusion of multiple myeloma, Waldenström macroglobulinemia, or other lymphoplasmacytic proliferative disorders.
8. Organ involvement: At least one organ affected (kidney, heart, liver, nervous system, gastrointestinal tract, lung, soft tissue) as per consensus guidelines.
9. Expected survival time ≥12 weeks.
10. Subjects must have adequate organ function, meeting all of the following laboratory criteria prior to enrollment:

    1. Complete blood count: Absolute neutrophil count (ANC) ≥1×10⁹/L; absolute lymphocyte count (ALC) ≥0.3×10⁹/L.
    2. Hemoglobin >60 g/L (no red blood cell [RBC] transfusion within 7 days prior to testing; use of recombinant human erythropoietin allowed).
    3. Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5× upper limit of normal (ULN); total serum bilirubin ≤1.5× ULN.
    4. Renal function: Creatinine clearance (CrCl) ≥30 mL/min as calculated by the Cockcroft-Gault formula.
    5. Coagulation function: Fibrinogen ≥1.0 g/L; activated partial thromboplastin time (APTT) ≤1.5× ULN; prothrombin time (PT) ≤1.5× ULN.
    6. Blood oxygen saturation >91%.
    7. Echocardiogram showing left ventricular ejection fraction (LVEF) ≥40%.
    8. Systolic blood pressure (SBP) ≥90 mmHg (oral vasopressor support allowed).
11. Subjects and their spouses agree to use effective contraceptive methods (tools or medications) from the time of signing the informed consent form until one year after CAR-T cell infusion.
12. Subjects voluntarily sign the informed consent form (ICF).

Exclusion Criteria:

1. Subjects who have received any of the following treatments prior to enrollment:

   1. Gene therapy before enrollment;
   2. Live vaccine within 4 weeks before enrollment;
   3. Other interventional clinical trial drugs within 12 weeks before leukapheresis.
2. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with detectable hepatitis B virus (HBV) DNA in peripheral blood; positive for hepatitis C virus (HCV) antibody with detectable HCV RNA in peripheral blood; positive for human immunodeficiency virus (HIV) antibody; positive for cytomegalovirus (CMV) DNA; positive for syphilis testing.
3. Use of therapeutic doses of corticosteroids (defined as prednisone or equivalent >20 mg/day) within 7 days before screening, though physiological replacement, topical, and inhaled steroids are permitted.
4. Presence of uncontrolled active infection within 7 days before peripheral blood mononuclear cell (PBMC) collection (excluding genitourinary system infections and upper respiratory tract infections <CTCAE Grade 2).
5. Receipt of any systemic therapy for AL amyloidosis within 14 days before PBMC collection.
6. Undergoing major surgery within 14 days before PBMC collection, or planning surgery within 2 weeks after study treatment (subjects planning local anesthesia surgery are eligible to participate).
7. Unresolved non-hematologic toxicity from prior therapy to baseline or ≤Grade 1 (per NCI-CTCAE v5.0, excluding alopecia and Grade 2 peripheral neuropathy).
8. Known life-threatening allergic reaction, hypersensitivity, or intolerance to cellular products or their components.
9. Subjects with suspected or confirmed symptoms of central nervous system (CNS) involvement by plasma cell tumors.
10. Bone marrow plasma cells >30% with clinical symptoms of multiple myeloma accompanied by osteolytic bone lesions.
11. Severe active cardiovascular disease with significant clinical symptoms despite treatment, including but not limited to unstable angina, myocardial infarction, and severe arrhythmia (excluding those with implanted implantable cardioverter-defibrillator [ICD] or pacemaker).
12. Subjects with bleeding or severe thrombosis symptoms as judged by the investigator, or with genetic/acquired bleeding and severe thrombosis conditions (including hemophilia, coagulopathy, thrombocytopenia, splenomegaly), or currently receiving thrombolytic or anticoagulant therapy.
13. Subjects with hypertension that cannot be controlled by medication.
14. Subjects who have received solid organ transplantation.
15. Subjects with a history of central nervous system disorders (e.g., cerebral aneurysm, epilepsy, stroke, dementia, psychosis) or consciousness impairment.
16. Subjects with unstable systemic diseases as judged by the investigator, including but not limited to severe liver, kidney, or metabolic diseases requiring medical treatment.
17. Diagnosis of malignancy other than multiple myeloma within 5 years before screening, excluding adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer post-radical surgery, or ductal carcinoma in situ of the breast post-radical surgery.
18. Participation in another interventional clinical trial within 1 month before signing the ICF.
19. Women who are pregnant, breastfeeding, or planning to become pregnant.
20. Subjects who do not agree to or have not completed the signing of the ICF.
21. Other conditions deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Achieving Hematologic VGPR or Better by Day 90 | From Eque-cel infusion to Day 90 post-infusion
  This measure assesses the effectiveness of Eque-cel CAR-T therapy by calculating the percentage of patients who achieve a Very Good Partial Response (VGPR) or better within 90 days post-infusion. Hematologic response indicates a significant reduction in AL amyloidosis blood markers, like abnormal light chains, based on international consensus guidelines. Blood samples are tested at Day 90 using lab methods such as serum free light chain (FLC) and protein electrophoresis (SPEP) to confirm VGPR, reflecting disease control in Mayo Stage IIIb patients.

SECONDARY OUTCOMES:
Complete Hematologic Response Rate (CHR) | From Eque-cel infusion to 24 months
  The proportion and time to achieving complete hematologic response as defined by the international consensus criteria for amyloidosis.
Major Organ Deterioration-Progression-Free Survival (MOD-PFS) | From the time of Eque-cel infusion up to 24 months
  This composite endpoint is defined as the time from randomization to the first occurrence of any of the following events (whichever comes first)：
  1. Death;
  2. Clinical manifestation of heart failure: defined as dyspnea at rest (for at least 3 consecutive days) solely due to amyloid cardiomyopathy, or the need for heart transplantation, left ventricular assist device (LVAD), or intra-aortic balloon pump (IABP);
  3. Clinical manifestation of renal failure: defined as progression to end-stage renal disease (requiring hemodialysis or kidney transplantation); hematologic progression as per consensus criteria: from CHR, any detectable monoclonal protein or abnormal free light chain ratio (ratio must double); from PR, a 50% increase in serum M protein to >0.5 g/dL or a 50% increase in urine M protein to >200 mg/day (measurable peak required); a 50% increase in free light chains to >100 mg/L.
Progression-Free Survival (PFS) | From the time of Eque-cel infusion up to 24 months
  Defined as the time from screening/enrollment to the first documentation of hematologic disease progression, organ (cardiac, renal, or hepatic) progression, or death from any cause (whichever occurs first), based on laboratory results and determined by international consensus criteria.
Organ Response Rate (OrRR) | From the time of Eque-cel infusion up to 24 months
  The proportion of patients with baseline organ involvement achieving a response in each respective organ within 24 months.
Overall Survival (OS) | From the time of Eque-cel infusion up to 24 months
  Defined as the time from screening/enrollment to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Liu peng, Professor, Study Chair — Fudan University

IPD SHARING:
Plan to Share IPD: No